CLINICAL TRIAL: NCT05385848
Title: Autologous Platelet-rich Plasma (PRP) Infusion to Improve Outcomes in Women With Ovarian Insufficiency: a Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Loh Jia Min Michelle, Principal Investigator, KK Women's and Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIRB 2022/2222
Record Dates: First submitted 2022-05-04; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Diminished Ovarian Reserve; Premature Ovarian Insufficiency; Fertility Issues; IVF
Keywords: Diminished Ovarian Reserve; Premature Ovarian Insufficiency; Poor Ovarian Reserve; Platelet-rich plasma; PRP; In Vitro Fertilisation (IVF); Fertility
MeSH Terms: conditions — Primary Ovarian Insufficiency; Infertility | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRP Injection Arm (Experimental): All patients recruited will come down to KKIVF Centre on Day 2-3 of the menstrual cycle to do blood tests (Anti-Mullerian Hormone (AMH)) and an ultrasound scan (Antral Follicular Count (AFC)). In the same menstrual cycle/month, autologous PRP injection will be done on Day 5-15 of the cycle.
  Patients will return to KKIVF Centre 1-3 months after the PRP injection on Day 2-3 of the menstrual cycle to repeat blood tests (AMH) and Ultrasound scan (AFC).
  IVF stimulation cycle as per KKIVF protocol will be started within 6 months from PRP injection. Patients will be followed up as per routine, with no more additional visits pertaining specifically to the study.
  Interventions: Procedure: Autologous Platelet-rich Plasma (PRP) Injection

INTERVENTIONS:
Procedure: Autologous Platelet-rich Plasma (PRP) Injection — PRP contains a high concentration of platelets which contains multiple vaso-active peptides and cytokines such as Vascular Endothelial Growth Factor (VEGF), Platelet-Derived Growth Factor (PDGF) and Sphingosine-1-phosphate. Many of these cytokines have been implicated in important roles in ovarian function, follicular genesis and oocyte maturation. Intraovarian autologous PRP infusion was recently introduced in the context of addressing ovarian insufficiency, with several studies showing an increase in ovarian function and promising ART outcomes. Possible mechanisms include anti-inflammatory and mitogenic potentials in this growth factor rich fraction contributing towards tissues regeneration. Through being involved in the cell regeneration cycle, autologous PRP potentially gives women with premature ovarian insufficiency (POI) or diminished ovarian insufficiency (DOR) hope in achieving a healthy genetically related offspring.

SUMMARY:
The investigators propose a pilot study to determine if autologous platelet-rich plasma (PRP) improves ovarian reserves and In-vitro fertilisation (IVF) outcomes in women with diminished ovarian reserve / premature ovarian insufficiency.

DETAILED DESCRIPTION:
Ovarian aging is a principal limiting factor for success in both spontaneous and assisted reproductive techniques (ART) conceptions. This results in diminished ovarian reserve (DOR) and premature ovarian insufficiency (POI), accounting for ~10% of IVF patients in Singapore and worldwide. Existing solutions include nutritional supplementations, high dose gonadotrophin usage, and experimental in-vitro activation with limited effectiveness, while donor oocyte programs or adoption do not provide a genetically related offspring. The substantial clinical burden and lack of effective treatments underscore the highly unmet need in this group of women.

Intraovarian autologous platelet-rich plasma (PRP) infusion was recently introduced in the context of addressing ovarian insufficiency, with several studies showing an increase in ovarian function and promising ART outcomes. Possible mechanism includes anti-inflammatory and mitogenic potentials in this growth factor rich fraction contributing towards tissues regeneration. Through being involved in the cell regeneration cycle, autologous PRP potentially gives women with POI/DOR a hope in achieving a healthy genetically related offspring. It however, still remains an experimental technique as there are very few small studies published till date, with no locally published data on its use.

The investigators propose a pilot study in KK Women's and Children's Hospital IVF (KKIVF) Centre to establish technical expertise, and to evaluate response to PRP to power a randomized controlled trial eventually. Primary outcomes are Anti-Mullerian Hormone (AMH), D2/3 Antral Follicle Count (AFC) and number of oocytes collected at stimulation. The secondary outcome will be clinical pregnancy and live birth rates. Thirty women with DOR/POI will be recruited over a 1 year period. The investigators hypothesize that PRP increases the overall pregnancy and live birth rates in these women.

ELIGIBILITY:
Inclusion criteria

* Diminished ovarian reserves AND/OR;
* Anti-Mullerian Hormone (AMH) 0.2-0.5ng/ml or
* At least 2 Follicle Stimulating Hormone (FSH) readings of >25 (mIU/L) or
* AFC < 5
* Poor Ovarian Response of <4 oocytes retrieved at a prior IVF stimulation cycle with gonadotrophin doses of 450u per day

Exclusion criteria

* Amenorrhea of > 1 years
* Medical conditions - Diabetes Mellitus, Hypertension, Collagen vascular diseases, Thyroid disease
* Patients presenting with anemia and thrombophilic disorders
* Inability to be monitored for at least 1 year at the treating centre
* Lack of suitable sperm for Intracytoplasmic Sperm Injection (ICSI) (eg. Azoospermia)

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only females will be recruited in this study.
Enrollment: 30 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change in ovarian reserves - Anti-Mullerian Hormone (AMH) | Baseline, and 4 to 12 weeks after PRP infusion
  Markers of ovarian reserve will be measured - Anti-Mullerian Hormone (AMH) levels on Day 2-3 of menses. Changes in ovarian reserve will be measured before and after the PRP infusion.
Change in ovarian reserves - Antral Follicular Count (AFC) | Baseline, and 4 to 12 weeks after PRP infusion
  Markers of ovarian reserve will be measured - Antral Follicular Count (AFC) on Day 2-3 of menses. Changes in ovarian reserve will be measured before and after the PRP infusion.

SECONDARY OUTCOMES:
Clinical pregnancy rates | Through study completion, an average of 10 months
  This is defined as the presence of fetal heartbeat or gestational sac at 6-9 weeks after fresh embryo transfer.
Live birth rates | Through study completion, an average of 10 months
  Live birth rates before and after 37 weeks of gestation will be one of the secondary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Loh, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No